CLINICAL TRIAL: NCT03935178
Title: A Single-Center, Blinded, Randomized Control Trial Evaluating Different Approaches to Evaluation of Right Ventricular Size and Function Using the Upper Valley Right Ventricle Algorithm and Novel Imaging Modalities
Brief Title: Evaluating Right Ventricular (RV) Size and Function Using the Upper Valley RV Algorithm and Novel Imaging Modalities
Acronym: UVRV
Status: Terminated | Type: Observational
Why Stopped: funding
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Eric S. Rothstein, Staff Physician, Heart and Vascular Center, Dartmouth-Hitchcock Medical Center
Other Study IDs: D19082 HVC 2019
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Hypertension; Valvular Heart Disease; Congenital Heart Disease; Congestive Heart Failure; Pulmonary Embolism; Acute Coronary Syndrome
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Valve Diseases; Heart Defects, Congenital; Heart Failure; Pulmonary Embolism; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Measuring Right Ventricular Size and Function — This study focuses on evaluating different approaches to evaluation of right ventricular size and function using the Upper Valley Right Ventricle Algorithm and novel imaging modalities

SUMMARY:
The primary purpose of this study is to evaluate the diagnostic performance of three methods for measuring right ventricular size and function including the Philips Novel RV quantification technologies (RV Heart Model volumetric analysis and Philips 2D strain) and the Upper Valley Right Ventricle Algorithm (UVRV) algorithm as compared to the gold standard of volumetric analysis via cardiac magnetic resonance imaging (CMR) in a broad patient population.

DETAILED DESCRIPTION:
This is a single-center, blinded, randomized control trial of patients 18-years or older that are undergoing CMR as a standard of care at Dartmouth-Hitchcock Medical Center in Lebanon, NH. After informed consent is obtained, subjects undergo a study-specific external, non-invasive echocardiogram utilizing a special RV focused protocol on the same day of their CMR as close to their scheduled CMR as possible to minimize wait time for consented patients. The echocardiogram takes approximately an additional 30 minutes of the subject's time.

De-identified echocardiogram images from each subject will be evaluated by experienced echocardiographers using three different methodologies (standard method, Phillips Novel technology and the newly developed UVRV algorithm). The methodologies will be compared with each other to determine sensitivity, specificity and accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patient age is over 18 years
* Patient is undergoing Cardiac MRI with sequences that permit biventricular volumetric analysis
* Patient is capable of giving informed consent
* The cardiac MRI images are of diagnostic quality to provide accurate RV and LV volumes

Exclusion Criteria:

- Patient unable to under echocardiogram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is for people who are18-years or older that are undergoing cardiac magnetic resonance imaging (CMR) as a standard of care at Dartmouth-Hitchcock Medical Center in Lebanon, NH.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Echocardiographic measurement - Right ventricular size | Echocardiographic measurements are taken on the same day as the scheduled CMR, as close to the scheduled CMR as possible, approximately 1 hour
  De-identified echocardiogram images from each subject will be evaluated by experienced echocardiographers using three (3) different methodologies. Specific evaluating MRI derived right ventricular volumes versus various echo approaches to grading right ventricular size.
Echocardiographic measurement - Right ventricular function | Echocardiographic measurements are taken on the same day as the scheduled CMR as possible, as close to the scheduled CMR, approximately 1 hour
  De-identified echocardiogram images from each subject will be evaluated by experienced echocardiographers using three (3) different methodologies.
Echocardiographic measurement - Right ventricular dysfunction severity | Echocardiographic measurements are taken on the same day as the scheduled CMR as possible, as close to the scheduled CMR, approximately 1 hour
  De-identified echocardiogram images from each subject will be evaluated by experienced echocardiographers using three (3) different methodologies. Severity reported as mild, moderate or severe)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Friedman, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant echocardiographic data that underlie the results reported in all publications will be shared after deidentification (text, tables, figures and appendices). The informed consent and study plan will also be shared following publication of the study results.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Information will be made available to researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Graham TP Jr, Bernard YD, Mellen BG, Celermajer D, Baumgartner H, Cetta F, Connolly HM, Davidson WR, Dellborg M, Foster E, Gersony WM, Gessner IH, Hurwitz RA, Kaemmerer H, Kugler JD, Murphy DJ, Noonan JA, Morris C, Perloff JK, Sanders SP, Sutherland JL. Long-term outcome in congenitally corrected transposition of the great arteries: a multi-institutional study. J Am Coll Cardiol. 2000 Jul;36(1):255-61. doi: 10.1016/s0735-1097(00)00682-3. PMID 10898443
- [Background] Chaowalit N, Durongpisitkul K, Krittayaphong R, Komoltri C, Jakrapanichakul D, Phrudprisan S. Echocardiography as a simple initial tool to assess right ventricular dimensions in patients with repaired tetralogy of Fallot before undergoing pulmonary valve replacement: comparison with cardiovascular magnetic resonance imaging. Echocardiography. 2012 Nov;29(10):1239-46. doi: 10.1111/j.1540-8175.2012.01766.x. Epub 2012 Jul 2. PMID 22748061
- [Background] Burgess MI, Mogulkoc N, Bright-Thomas RJ, Bishop P, Egan JJ, Ray SG. Comparison of echocardiographic markers of right ventricular function in determining prognosis in chronic pulmonary disease. J Am Soc Echocardiogr. 2002 Jun;15(6):633-9. doi: 10.1067/mje.2002.118526. PMID 12050605
- [Background] D'Alonzo GE, Barst RJ, Ayres SM, Bergofsky EH, Brundage BH, Detre KM, Fishman AP, Goldring RM, Groves BM, Kernis JT, et al. Survival in patients with primary pulmonary hypertension. Results from a national prospective registry. Ann Intern Med. 1991 Sep 1;115(5):343-9. doi: 10.7326/0003-4819-115-5-343. PMID 1863023
- [Background] de Groote P, Millaire A, Foucher-Hossein C, Nugue O, Marchandise X, Ducloux G, Lablanche JM. Right ventricular ejection fraction is an independent predictor of survival in patients with moderate heart failure. J Am Coll Cardiol. 1998 Oct;32(4):948-54. doi: 10.1016/s0735-1097(98)00337-4. PMID 9768716
- [Background] Dursunoglu N, Dursunoglu D, Yildiz AI, Rota S. Evaluation of cardiac biomarkers and right ventricular dysfunction in patients with acute pulmonary embolism. Anatol J Cardiol. 2016 Apr;16(4):276-82. doi: 10.5152/akd.2014.5828. Epub 2014 Dec 31. PMID 26645262
- [Background] Mehta SR, Eikelboom JW, Natarajan MK, Diaz R, Yi C, Gibbons RJ, Yusuf S. Impact of right ventricular involvement on mortality and morbidity in patients with inferior myocardial infarction. J Am Coll Cardiol. 2001 Jan;37(1):37-43. doi: 10.1016/s0735-1097(00)01089-5. PMID 11153770
- [Background] Zehender M, Kasper W, Kauder E, Geibel A, Schonthaler M, Olschewski M, Just H. Eligibility for and benefit of thrombolytic therapy in inferior myocardial infarction: focus on the prognostic importance of right ventricular infarction. J Am Coll Cardiol. 1994 Aug;24(2):362-9. doi: 10.1016/0735-1097(94)90289-5. PMID 8034869
- [Background] Anavekar NS, Gerson D, Skali H, Kwong RY, Yucel EK, Solomon SD. Two-dimensional assessment of right ventricular function: an echocardiographic-MRI correlative study. Echocardiography. 2007 May;24(5):452-6. doi: 10.1111/j.1540-8175.2007.00424.x. PMID 17456062
- [Background] Bleeker GB, Steendijk P, Holman ER, Yu CM, Breithardt OA, Kaandorp TA, Schalij MJ, van der Wall EE, Nihoyannopoulos P, Bax JJ. Assessing right ventricular function: the role of echocardiography and complementary technologies. Heart. 2006 Apr;92 Suppl 1(Suppl 1):i19-26. doi: 10.1136/hrt.2005.082503. No abstract available. PMID 16543597
- [Background] Helbing WA. Right ventricular function: the comeback of echocardiography? Eur J Echocardiogr. 2004 Mar;5(2):99-101. doi: 10.1016/j.euje.2003.12.001. No abstract available. PMID 15036018
- [Background] Jorstig S, Waldenborg M, Liden M, Thunberg P. Right ventricular ejection fraction measurements using two-dimensional transthoracic echocardiography by applying an ellipsoid model. Cardiovasc Ultrasound. 2017 Mar 7;15(1):4. doi: 10.1186/s12947-017-0096-5. PMID 28270161
- [Background] Zornoff LA, Skali H, Pfeffer MA, St John Sutton M, Rouleau JL, Lamas GA, Plappert T, Rouleau JR, Moye LA, Lewis SJ, Braunwald E, Solomon SD; SAVE Investigators. Right ventricular dysfunction and risk of heart failure and mortality after myocardial infarction. J Am Coll Cardiol. 2002 May 1;39(9):1450-5. doi: 10.1016/s0735-1097(02)01804-1. PMID 11985906
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] Kjaergaard J, Petersen CL, Kjaer A, Schaadt BK, Oh JK, Hassager C. Evaluation of right ventricular volume and function by 2D and 3D echocardiography compared to MRI. Eur J Echocardiogr. 2006 Dec;7(6):430-8. doi: 10.1016/j.euje.2005.10.009. Epub 2005 Dec 9. PMID 16338173
- [Background] Pfluger HB, Maeder MT, LaGerche A, Taylor AJ. One- and two-dimensional estimation of right and left ventricular size and function-comparison with cardiac magnetic resonance imaging volumetric analysis. Heart Lung Circ. 2010 Sep;19(9):541-8. doi: 10.1016/j.hlc.2010.03.003. Epub 2010 Apr 24. PMID 20457009
- [Background] DeLong ER, DeLong DM, Clarke-Pearson DL. Comparing the areas under two or more correlated receiver operating characteristic curves: a nonparametric approach. Biometrics. 1988 Sep;44(3):837-45. PMID 3203132
- [Background] Ahmad H, Mor-Avi V, Lang RM, Nesser HJ, Weinert L, Tsang W, Steringer-Mascherbauer R, Niel J, Salgo IS, Sugeng L. Assessment of right ventricular function using echocardiographic speckle tracking of the tricuspid annular motion: comparison with cardiac magnetic resonance. Echocardiography. 2012;29(1):19-24. doi: 10.1111/j.1540-8175.2011.01519.x. Epub 2011 Oct 4. PMID 21967480
- [Background] Giusca S, Dambrauskaite V, Scheurwegs C, D'hooge J, Claus P, Herbots L, Magro M, Rademakers F, Meyns B, Delcroix M, Voigt JU. Deformation imaging describes right ventricular function better than longitudinal displacement of the tricuspid ring. Heart. 2010 Feb;96(4):281-8. doi: 10.1136/hrt.2009.171728. Epub 2009 Aug 30. PMID 19720609
- [Background] Guendouz S, Rappeneau S, Nahum J, Dubois-Rande JL, Gueret P, Monin JL, Lim P, Adnot S, Hittinger L, Damy T. Prognostic significance and normal values of 2D strain to assess right ventricular systolic function in chronic heart failure. Circ J. 2012;76(1):127-36. doi: 10.1253/circj.cj-11-0778. Epub 2011 Oct 27. PMID 22033348
- [Background] Hardegree EL, Sachdev A, Villarraga HR, Frantz RP, McGoon MD, Kushwaha SS, Hsiao JF, McCully RB, Oh JK, Pellikka PA, Kane GC. Role of serial quantitative assessment of right ventricular function by strain in pulmonary arterial hypertension. Am J Cardiol. 2013 Jan 1;111(1):143-8. doi: 10.1016/j.amjcard.2012.08.061. Epub 2012 Oct 23. PMID 23102474
- [Background] Maffessanti F, Gripari P, Tamborini G, Muratori M, Fusini L, Alamanni F, Zanobini M, Fiorentini C, Caiani EG, Pepi M. Evaluation of right ventricular systolic function after mitral valve repair: a two-dimensional Doppler, speckle-tracking, and three-dimensional echocardiographic study. J Am Soc Echocardiogr. 2012 Jul;25(7):701-8. doi: 10.1016/j.echo.2012.03.017. Epub 2012 Apr 25. PMID 22542273
- [Background] Shimada YJ, Shiota M, Siegel RJ, Shiota T. Accuracy of right ventricular volumes and function determined by three-dimensional echocardiography in comparison with magnetic resonance imaging: a meta-analysis study. J Am Soc Echocardiogr. 2010 Sep;23(9):943-53. doi: 10.1016/j.echo.2010.06.029. PMID 20797527
- [Background] Petersen SE, Aung N, Sanghvi MM, Zemrak F, Fung K, Paiva JM, Francis JM, Khanji MY, Lukaschuk E, Lee AM, Carapella V, Kim YJ, Leeson P, Piechnik SK, Neubauer S. Reference ranges for cardiac structure and function using cardiovascular magnetic resonance (CMR) in Caucasians from the UK Biobank population cohort. J Cardiovasc Magn Reson. 2017 Feb 3;19(1):18. doi: 10.1186/s12968-017-0327-9. PMID 28178995